CLINICAL TRIAL: NCT01206894
Title: Pre-Operative Assessment of Chest Wall Invasion in Non-Small Cell Lung Cancer (NSCLC)Using Pre-Operative, Surgeon Performed Ultrasound
Brief Title: Pre-Operative Assessment of Chest Wall Invasion in NSCLC Using Pre-Operative, Surgeon Performed Ultrasound
Acronym: CT0010
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE 10.119
Record Dates: First submitted 2010-09-14; First posted 2010-09-22 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung cancer; chest wall invasion; transthoracic ultrasound
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Transthoracic Ultrasound — 1 transthoracic ultrasound will be performed the evening before the thoracic surgery
  Other Names: Chest wall invasion

SUMMARY:
Non-Small Cell Lung Cancer (75% of lung cancer) is associated with involvement of the parietal pleura and or chest wall (soft tissue and/or bone) in 5-8% of patients. Invasion of the chest wall increases the T staging in the Tumor, Node, Mestasis (TNM) classification system of lung cancer to a T3 and is associated with decreased survival and more extensive operative procedures. The reported 5-year survival for patients with T2 tumors is 58% compared to 38% in patients with T3 lesions. The American college of Chest Physician has still not identified the best tool to assess chest wall invasion by lung cancer, CT-Scan being used by physicians for this assessment. In some studies, CT scan has been shown to have a sensitivity ranging from 42 % to 68 % in assessing chest wall invasion, and a specificity ranging from 66 % to 100 %.

Trans-thoracic Ultrasound (US) has the capacity of allowing for dynamic real-time imaging of the pulmonary lesion and the chest wall. Therefore, US has the potential to allow for the appreciation of subtle findings related to the movement of the lesion and lung over the chest wall. Hence, US might be an accurate tool to assess chest wall invasion by lung cancer; thus improving pre-operative diagnosis, staging and operative planning of patient with chest wall invasion.

However US is not currently utilized in the pre-operative assessment of patients with lung cancer invading the pleura and chest wall, and has not been extensively studied.

In some rare studies evaluating the accuracy of US, results have shown a sensitivity ranging from 89% to 100% and a specificity ranging from 95% to 98% for US detecting chest wall invasion by lung cancer. However those studies got criticized. Bandi et al study, got criticized by the fact that the operators in the study were experienced interventional pulmonologists who perform hundreds of thoracic and endoscopic ultrasound per year. Nobuo et al study took place in 1993, since when the device of US has evolved, the investigators can not apply with certainty the findings of this study.

Consequently, there is a need to conduct a study to evaluate the accuracy of US to assess chest wall invasion by lung cancer.

In this prospective study the investigators will assess the accuracy of US, and then compare it to the accuracy of the CT-Scan

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral pulmonary nodules abutting the visceral pleura on pre-operative CT scan of the chest and who are booked for surgery.

Exclusion Criteria:

* Inability to consent for the study.
* Patients less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the accuracy of real-time chest ultrasonographic in assessing chest wall invasion compared to Ultrasound | 3-6 months
  Sensitivity, specificity will be calculated for US and CT scan for assessing chest wall invasion.

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Tahiri M, Khereba M, Thiffault V, Ferraro P, Duranceau A, Martin J, Liberman M. Preoperative assessment of chest wall invasion in non-small cell lung cancer using surgeon-performed ultrasound. Ann Thorac Surg. 2014 Sep;98(3):984-9. doi: 10.1016/j.athoracsur.2014.04.111. Epub 2014 Jul 16. PMID 25038014